CLINICAL TRIAL: NCT06826963
Title: The Role of Eccentric Exercise in the Older Sarcopenic Population with Heart Failure: a Feasibility and Efficacy Study Protocol
Brief Title: Feasibility and Effectiveness of Eccentric Exercise in Sarcopenic Older Adults with Heart Failure: a Pilot Study
Acronym: ECLYPSE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Valentina Muollo, Ph.D., PhD, Universita di Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prot. n. 45282 date 13/08/2024; CUP B43C22000450006 (Other Grant/Funding Number: Interconnected Nord-Est Innovation Ecosystem (iNEST) (Verona, Verona, IT))
Record Dates: First submitted 2025-01-22; First posted 2025-02-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure with Preserved Ejection Fraction (HFPEF); Heart Failure with Reduced Ejection Fraction; Sarcopenia in Elderly; Sarcopenic Obesity
Keywords: eccentric exercise; older adults; heart failure; sarcopenia; sarcopenic obesity; muscle strength; muscle mass; exercise intervention; aging
MeSH Terms: conditions — Heart Failure; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Older adults with sarcopenia and heart failure (Experimental): Men and women aged 65 to 85 years, with stable heart failure (HF) (either preserved left ventricular ejection fraction (≥50%) or reduced ejection fraction (≤40%)). Eligibility requires classification as New York Heart Association (NYHA) class 1, 2, or 3, and meeting the diagnostic criteria for sarcopenia or sarcopenic obesity. Sarcopenic patients are classified by skeletal muscle mass index (kg/m²): class I (males ≤10.75, females ≤6.75) and class II (males ≤8.50, females ≤5.75). For sarcopenic obesity, the classifications are: class I (males 31.3-37%, females 22.1-27.6%) and class II (males <31.5%, females <22.1%). This arm will participate in a supervised eccentric cycling training program for three months. The intervention will include two training sessions per week in the first month, increasing to three sessions per week in the following two months.
  Interventions: Other: Aerobic eccentric intervention

INTERVENTIONS:
Other: Aerobic eccentric intervention — This arm will participate in a supervised eccentric cycling training program for three months. The intervention will include two training sessions per week in the first month, increasing to three sessions per week in the following two months. Each session will consist of a warm-up (5 minutes), a main training phase (20-30 minutes), and a cool-down (5-10 minutes). The intensity of training will be gradually adjusted to maintain a perceived exertion rating (RPE) between light and moderate with a target heart rate zone (57-76% of HRmax). Pre- and post-training assessments will evaluate physical function through several tests, body composition and anthropometric indices, muscle strength of upper and lower limbs, questionnaires related to the overall health improvement. Finally, participants will also be monitored for daily physical activity through wearable sensors to track mobility and autonomy.

SUMMARY:
This study is designed to evaluate the safety, feasibility, and effectiveness of a 12-week eccentric exercise program for older adults with sarcopenia (muscle loss) or sarcopenic obesity and chronic heart failure (HF). The program aims to improve physical performance, muscle strength, and overall health without causing excessive strain on participants. Eccentric exercise has shown potential benefits for improving muscle function, and this study will help determine if it is a safe and effective option for individuals with heart failure and muscle loss.

Study Goals: The primary aim of this study is to test the feasibility and effectiveness of an eccentric exercise program for older adults with sarcopenia and CHF. The study will monitor physical performance, adherence to the program, and participants' ability to tolerate the exercise, as well as any impact on heart and muscle health.

Study Population: A screening visit will be scheduled to determine if individuals meet the criteria to participate in the study. During this visit, a detailed assessment will be made, and if eligible, participants will sign an informed consent form.

This study will assess whether a 12-week eccentric exercise program can help improve muscle strength, cardiovascular health, and overall physical performance in individuals with HF and sarcopenia. The program will involve exercising on an eccentric bike, which is designed to reduce strain on the heart while providing effective muscle strengthening benefits.

The study will use several physical performance tests to assess the impact of the exercise program, including:

1. Short Physical Performance Battery (SPPB): Evaluates mobility and strength.
2. 6-Minute Walk Test (6MWT): Measures cardiovascular fitness.
3. Handgrip Strength and Leg Strength Tests: Assess upper and lower body muscle strength.
4. Additionally, body composition will be evaluated using tools such as DXA scans and bioelectrical impedance analysis (BIA) to measure muscle mass, fat, and overall health status. The program's adherence and tolerance will be carefully monitored by measuring session completion, intensity, and participant feedback.

Primary Outcomes

Feasibility Measures:

1. Recruitment and Completion Rate: The ratio of participants recruited to those who successfully complete the study, including post-intervention assessments.
2. Session Attendance: The number of training sessions attended out of the total planned sessions.
3. Adherence to Training Volume: The number of prescribed exercises completed by participants compared to the total planned.
4. Program Tolerance: Evaluated by comparing the Rate of Perceived Exertion (RPE) during sessions to the target RPE.

To be considered feasible, the study must meet these criteria: Recruitment >50%, Follow-up loss <20%, Median attendance at training sessions >80%, Median adherence to prescribed volume >75%, Tolerance to RPE >70%.

Secondary Outcomes

Effectiveness Measures:

1. SARC-F: A tool for identifying individuals at risk of sarcopenia, based on self-reported issues like weakness and difficulty walking.
2. Mini Nutritional Assessment (MNA): Evaluates nutritional status to rule out malnutrition, which could affect training outcomes.
3. Mini Mental State Examination (MMSE): Assesses cognitive function.
4. Minnesota Living with Heart Failure Questionnaire: Evaluates how heart failure affects daily life.
5. International Physical Activity Questionnaire (IPAQ): Measures physical activity levels at baseline.

In addition to the physical performance tests mentioned, the study will assess muscle mass and fat distribution using DXA scans and BIA, providing a comprehensive view of body composition. Finally, the feasibility of remotely monitoring patients' physical activity to determine the impact of the intervention on their daily lives, specifically in terms of mobility and autonomy is assessed. To this end, patients will be asked to wear a set of five sensors (two on the ankles, two on the wrists, and one on the waist) for at least four days. The Axivity AX6 sensors, chosen for their light weight and long battery life, will collect data used to monitor time spent moving, sitting, and lying down, as well as to assess the quality of the recorded movements.

DETAILED DESCRIPTION:
Training protocol overview Familiarization Phase Before starting the actual training program, patients will undergo a familiarization phase to allow them to adjust to the eccentric cycling equipment and understand the intensity of the exercises. This phase is critical for ensuring safety and optimizing adherence to the program.

Duration of Familiarization:

The familiarization phase will last for two weeks. The first week (sessions 4 and 5, conducted within the same week after medical screening and body composition testing) will focus on achieving an intensity that is perceived as "very light" (RPE 8-9) and maintaining it for 5-10 minutes.

The second week will aim for a light (RPE 10-11) to slightly heavy (RPE 10-13) intensity.

Muscle Pain Monitoring:

At the beginning and end of each familiarization session, patients will be asked to rate their muscle pain using the Visual Analog Scale (VAS) (0-10), where 0 represents no pain and 10 indicates unbearable pain. This ensures that any discomfort is monitored and managed appropriately, reducing the risk of muscle injury and enhancing adherence to the program.

Purpose of Familiarization:

This phase helps patients adapt to eccentric training, preventing unnecessary muscle damage and ensuring they are comfortable with the equipment and the level of exertion. It also serves to acclimatize the patients to the specific eccentric muscle contractions involved in the cycling exercise.

Exercise Prescription Trained kinesiologists will supervise the eccentric cycling sessions. Monitoring and adjusting exercise intensity based on heart rate (HR) and Rate of Perceived Exertion (RPE) will be central to ensuring safety and effectiveness throughout the intervention.

Intensity Monitoring: For participants on beta-blockers, maximum heart rate (HRmax) will be estimated using the formula: HRmax = 164 - (0.7 × age). For participants not on beta-blockers, HRmax will be calculated using: HRmax = 211 - (0.64 × age).

The HR and RPE will be continuously monitored to ensure participants are training within the prescribed intensity zones.

Target Intensity: The training intensity will be kept between light (57-64% of HRmax) and moderate/slightly heavy (64-76% of HRmax) levels. These ranges correspond to RPE values of approximately 10-14.

The intensity will vary within the session, with three different workloads: Light: RPE ~10, Moderate: RPE ~12, Slightly Heavy: RPE ~14

Session Structure: Each training session will be divided into three parts:

1. Warm-Up (5 minutes): Low-intensity cycling to prepare the body.
2. Main Training (20-30 minutes): The main part of the session will focus on eccentric cycling at varying intensities. The patients will alternate between light, moderate, and slightly heavy intensities, maintaining the prescribed intensity range (RPE ~10-14).
3. Cool-Down (5-10 minutes): Gradual reduction in intensity to aid in recovery. Progressive Training Plan: Week 1-4 (Adaptation Phase): Patients will train twice a week, with an emphasis on familiarizing themselves with the bike and adjusting to the intensity ranges.

The duration of the central training phase will start at 20 minutes. Week 5-8 (Strengthening Phase): Training frequency will increase to three times per week. The duration of the central phase will increase progressively to 30 minutes. The intensity will gradually rise within the prescribed target range, increasing as the patients adapt.

Week 9-12 (Maximal Tolerable Load Phase): The frequency remains three times a week. The intensity will reach the higher end of the prescribed range, with patients performing the eccentric cycling at near-maximal intensities (RPE 14-15). Adjustments Every Two Weeks: Every two weeks, the workload will be reassessed and adjusted to ensure the target RPE is achieved and maintained. This will ensure continued progression and avoid plateauing.

Pedaling Frequency: Participants will be instructed to maintain a pedal cadence of 60 RPM (revolutions per minute) for each session. This will be a consistent cadence for the entire training phase.

ELIGIBILITY:
Participants must meet all of the following criteria:

* Age 65 to 85 years
* Diagnosed with stable heart failure (HF), defined as:
* Preserved left ventricular ejection fraction (≥50%) or
* Reduced ejection fraction (≤40%)
* Classified as New York Heart Association (NYHA) class 1, 2, or 3
* Meet the diagnostic criteria for sarcopenia or sarcopenic obesity:
* Sarcopenia: Impaired muscle strength with the Five-repetition chair stand test time >15 seconds (normal weight) or >17 seconds (patients with obesity)
* Reduced muscle mass according to the European Working Group on Sarcopenia (EWGSOP) or Sarcopenic Obesity: Based on the European Society for Clinical Nutrition and Metabolism (ESPEN) and the European Association for the Study of Obesity (EASO).
* For EWGSOP:

Sarcopenia as Class I: Skeletal muscle mass index (kg/m²)

* Males: ≤10.75 kg/m²
* Females: ≤6.75 kg/m²
* For EWGSOP:

Sarcopenia as Class II: Skeletal muscle mass index (kg/m²)

* Males: ≤8.50 kg/m²
* Females: ≤5.75 kg/m²
* For ESPEN-EASO:

Obesity: waist circumference calculated in centimeters (cm)

* Males: ≥102 cm
* Females: ≥ 88 cm Sarcopenia as Class I: Skeletal muscle index as a percentage of body weight (%)
* Males: 31.3-37%
* Females: 22.1-27.6%

Sarcopenia as Class II:

* Males: <31.5%
* Females: <22.1%

Exclusion Criteria:

Participants will be excluded if they meet any of the following conditions:

* Severe obstructive heart disease
* Aortic valve stenosis
* Severe arrhythmias identified during initial stress testing
* Intracavitary thrombosis
* Severe pulmonary hypertension (>70 mmHg)
* History of venous thromboembolism within the previous three months
* History of heart transplantation
* Medical conditions that significantly limit functional capacity beyond the impact of HF

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment and Retention Rate | Recruitment and retention will be assessed at baseline and week 12.
  The feasibility of implementing a three-month eccentric cycling training program will be assessed using the following individual measures: Recruitment and Retention Rate: % of enrolled participants who complete post-intervention assessments. (Units of measures: Percentage [%]) Criteria for Feasibility: • Recruitment>50%
Session Attendance | Session attendance will be monitored weekly, with a final assessment at week 12.
  The feasibility of implementing a three-month eccentric cycling training program will be assessed using the following individual measure: Session Attendance - Median number of training sessions attended relative to the total planned sessions. (Units of measures: Percentage [%]) Median session attendance>80%
Adherence to Training Volume | Adherence, will be monitored weekly, with a final assessment at week 12.
  The feasibility of implementing a three-month eccentric cycling training program will be assessed using the following individual measures: Adherence to Training Volume - Median percentage of prescribed exercises completed relative to the total planned. (Units of measures: Percentage [%])
  Criteria for Feasibility:
  • Median session attendance>80%
Program Tolerance | Program tolerance will be monitored weekly, with a final assessment at week 12.
  The feasibility of implementing a three-month eccentric cycling training program will be assessed using the following individual measure: Program Tolerance - Proportion of participants achieving the target Rate of Perceived Exertion (RPE) during sessions. (Units of measures: Percentage [%])

SECONDARY OUTCOMES:
SARC-F questionnaire | Pre and after 12 weeks
  score 0-10; The SARC-F questionnaire is a simple and widely used screening tool for sarcopenia, a condition characterized by the loss of muscle mass, strength, and function, often associated with aging and certain diseases.
MNA questionnaire | Pre and after 12 weeks
  The Mini Nutritional Assessment (MNA) is a validated screening tool designed to assess the nutritional status of older adults (aged 65 and above) and identify those at risk of malnutrition.
  (score 0-30)
MMSE questionnaire | Only at PRE test
  The Mini-Mental State Examination (MMSE) is a widely used cognitive screening tool designed to assess an individual's mental status and detect cognitive impairment, such as in dementia or mild cognitive impairment (MCI). (score 0-30).
Minnesota Living with HF Questionnaire | Pre and after 12 weeks
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a validated patient-reported outcome measure designed to assess the impact of heart failure (HF) on an individual's quality of life (QoL). It is widely used in clinical practice and research to evaluate the severity of symptoms, functional limitations, and emotional well-being in patients with heart failure (score 0-105).
Physical Activity Level (IPAQ) | Only at PRE.
  The International Physical Activity Questionnaire (IPAQ) is a widely used self-reported tool designed to assess physical activity levels in adults. It was developed by the World Health Organization (WHO) to provide a standardized method for evaluating physical activity across different countries and cultures. The IPAQ is commonly used in both research and public health settings to assess activity levels and promote physical activity.
  Total Physical Activity Score = Sum of the activity frequency (days per week) multiplied by the duration (minutes per day) for each activity intensity (vigorous, moderate, walking).
  The score is then categorized based on the thresholds above to identify low, moderate, or high activity levels.
Weight | Pre and after 12 weeks
  Measured by a scale. Values collected in kg.
Height | Only at PRE.
  Height measured by stadiometer. Values collected in meters (m).
Body Mass Index | Pre and after 12 weeks
  Body Mass Index (BMI) is a simple and widely used tool to assess body weight relative to height and categorize individuals into various weight status groups. While it does not directly measure body fat percentage, BMI is used as a general indicator of whether a person has a healthy weight for a given height. It is particularly useful for population-level assessments and as a quick screening tool in clinical settings. Calculated as weight (kg)/height² (m²), kg/m².
Waist circumference | Pre and after 12 weeks
  Waist circumference is a simple and widely used measure of abdominal fat. It is particularly important in assessing the risk of metabolic and cardiovascular diseases, as abdominal fat (specifically visceral fat) is associated with higher risks of conditions such as type 2 diabetes, hypertension, and heart disease.
  Measure in centimeters (cm).
Hip circumference | Pre and after 12 weeks
  Hip circumference is the measurement of the circumference around the widest part of the hips and buttocks, typically measured at the level of the greater trochanters (the bony prominence on the outer side of the hip).
  Measure in centimeters (cm).
Calf circumference | Pre and after 12 weeks
  Calf circumference is a simple measurement of the circumference around the widest part of the lower leg, specifically the gastrocnemius muscle area. It is often used in clinical and research settings to assess nutritional status, muscle mass, and vascular health, especially in individuals who may have muscle wasting or vascular conditions.
  Smaller calf circumference is often a marker of frailty and sarcopenia in older adults, which is linked to reduced physical function, increased risk of falls, and reduced mobility.
  Record the measurement: Measure in centimeters (cm).
Muscle mass | Pre and after 12 weeks
  Muscle Mass will be measured through a Dual-Energy X-ray Absorptiometry (DEXA). A DEXA scan is a highly accurate and widely used imaging technique primarily used to measure bone mineral density (BMD), but it can also provide detailed information about body composition, including muscle mass, fat mass, and bone mass. DEXA scans are commonly used in both clinical and research settings to assess muscle mass, fat distribution, and bone health.
  Values in kg.
Fat Mass | Pre and after 12 weeks
  Fat Mass will be measured through a Dual-Energy X-ray Absorptiometry (DEXA). A DEXA scan is a highly accurate and widely used imaging technique primarily used to measure bone mineral density (BMD), but it can also provide detailed information about body composition, including muscle mass, fat mass, and bone mass. DEXA scans are commonly used in both clinical and research settings to assess muscle mass, fat distribution, and bone health. Values in kg/%.
Bone Density | Pre and after 12 weeks
  Bone Density will be measured through a Dual-Energy X-ray Absorptiometry (DEXA). A DEXA scan is a highly accurate and widely used imaging technique primarily used to measure bone mineral density (BMD), but it can also provide detailed information about body composition, including muscle mass, fat mass, and bone mass. DEXA scans are commonly used in both clinical and research settings to assess muscle mass, fat distribution, and bone health. Values in g/cm².
Short Physical Performance Battery | Pre and after 12 weeks
  The Short Physical Performance Battery (SPPB) is a widely used clinical assessment tool designed to measure lower extremity function and physical performance in older adults. It is particularly useful for identifying early signs of frailty, functional decline, and mobility issues. The SPPB is a brief and reliable tool that evaluates multiple aspects of physical function through a series of simple tasks. The SPPB consists of three main tests: Gait Speed Test, Balance Test and Chair Stand Test.
  The SPPB provides a total score based on the performance of each test.
  The total score ranges from 0 to 12 points, with higher scores indicating better overall physical performance.
Six Minute Walking Test | Pre and after 12 weeks
  The 6-Minute Walk Test (6MWT) is a simple, widely used functional exercise test that measures an individual's endurance, aerobic capacity, and physical fitness. It is commonly used in clinical and research settings to assess the functional status and exercise tolerance of individuals. The person is instructed to walk continuously without running or stopping (unless necessary), and to pace themselves at a speed they feel comfortable with. The total distance walked in meters (m) is recorded at the end of the 6 minutes.
Ten Meter Walking Speed | Pre and after 12 weeks
  The Ten-Meter Walking Speed Test (10mWT) is a commonly used simple and reliable test to assess gait speed and walking ability in individuals, particularly older adults and those with health conditions affecting mobility. It provides valuable information about an individual's functional mobility and is often used in clinical and research settings to assess frailty, cognitive function, and the risk of falls. The subject is instructed to walk at their normal, comfortable pace over the 10-meter course. This test is performed without running and with the individual walking continuously from one end to the other.
  The time taken to cover the 10 meters is recorded, and the result is expressed in seconds (s) which can be used to assess walking speed in m/s.
HandGrip | Pre and after 12 weeks
  The Handgrip Strength Test is a simple and widely used measure of muscle strength, specifically the strength of the hand and forearm muscles. It is commonly used in clinical and research settings to assess overall muscle function, health, and frailty, particularly in older adults or individuals with conditions that may affect muscle strength and physical performance.
  The subject is asked to squeeze a handgrip dynamometer (a device designed to measure grip strength) as hard as possible for a few seconds for three attempts. The maximum force applied during the squeeze is recorded in kilograms (kg).
Isometric Force | Pre and after 12 weeks
  Isometric force testing with a Cybex dynamometer provides precise measurements of muscle strength, which are important for assessing an individual's functional ability, recovery, and rehabilitation progress.
  In this study, the subjects will perform maximal isometric contractions with the knee angle at 90 degrees. Two tests will be performed, separated by 2 minutes of recovery. The value will be expressed in Newton x Metre (Nm).
Isokinetic Force | Pre and after 12 weeks
  Isokinetic Force refers to the force exerted by a muscle during an isokinetic movement, where the velocity of the joint motion is kept constant throughout the range of motion. Isokinetic testing is often used to assess muscle strength, endurance, and power under controlled conditions.
  Isokinetic refers to a type of muscle contraction where the velocity of movement (the speed at which the limb moves) is kept constant by the testing equipment, regardless of the force the muscle is generating.
  This is achieved using isokinetic dynamometers, which can measure and control the speed of joint movement during the test (e.g., Cybex). These devices adjust resistance based on the muscle's output, ensuring that the joint velocity remains the same.
  In this study, the participants will perform two familiarization contractions and three evaluation contractions, both in extension and flexion, at the following speeds: 60, 90, 150, 180, and 210 °/s.
  The values will be recorded in Newton x Metre (Nm)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Verona, Italy